CLINICAL TRIAL: NCT03844230
Title: Role of Sweet Taste Signaling in Glucose Regulation
Brief Title: Role of Sweetness in Glucose Regulation
Acronym: STS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19294
Record Dates: First submitted 2019-01-29; First posted 2019-02-18 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: sweeteners; glucose metabolism; taste receptors; sucralose
MeSH Terms: conditions — Obesity | interventions — Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhibition Group (Other): Randomly selected habitual and non habitual LCS consumers will be assessed on three different oral glucose tolerance test conditions (i.e. Control - Inhibition, Experimental I- Inhibition, Experimental II- Inhibition). A separate visit will evaluate their sweet taste perception and preferences (Sensory evaluation).
  Interventions: Other: Control - Inhibition; Other: Experimental I- Inhibition; Other: Experimental II- Inhibition; Other: Sensory Evaluation
- Stimulation Group (Other): Randomly selected habitual and non habitual LCS consumers will be assessed on three different oral glucose tolerance test conditions (i.e. Control - Stimulation, Experimental I- Stimulation, Experimental II -Stimulation). A separate visit will evaluate their sweet taste perception and preferences (Sensory evaluation).
  Interventions: Other: Control- Stimulation; Other: Experimental I- Stimulation; Other: Experimental II- Stimulation; Other: Sensory Evaluation

INTERVENTIONS:
Other: Control - Inhibition — Taste and spit up water 10 minutes before drinking a glucose load
  Arms: Inhibition Group
Other: Experimental I- Inhibition — Taste and spit up water 10 minutes before drinking a glucose load mixed with lactisole
  Arms: Inhibition Group
Other: Experimental II- Inhibition — Taste and spit up sucralose 10 minutes before drinking a glucose load mixed with lactisole
  Arms: Inhibition Group
Other: Control- Stimulation — Taste and spit up water 10 minutes before drinking a glucose load
  Arms: Stimulation Group
Other: Experimental I- Stimulation — Taste and spit up sucralose 10 minutes before drinking a glucose load
  Arms: Stimulation Group
Other: Experimental II- Stimulation — Drink sucralose 10 minutes before drinking a glucose load
  Arms: Stimulation Group
Other: Sensory Evaluation — Taste different solutions to evaluate sweet taste preference, suprathreshold intensity and detection threshold

SUMMARY:
Data from several studies show that consuming a diet high in low-calorie sweeteners (LCS), mainly in diet sodas, is linked to the same metabolic disorders as consuming a diet high in added sugars, including an increased risk of developing type 2 diabetes. Sweet taste receptors, once thought to be unique to the mouth, have now been discovered in other parts of the body, including the intestine and the pancreas, where they play a role in blood sugar control. These newly identified receptors provide new avenues to explore how LCS may affect metabolism and health. This project is designed to examine the role of sweet taste signaling, both in the mouth and in the gut, on blood sugar control and how habitual consumption of LCS may affect sweet taste signaling and metabolism in people with obesity.

DETAILED DESCRIPTION:
The overall goal of this research is to assess the role of oral and gut sweetness signaling in postprandial glucose metabolism and to determine how acute and chronic low-calorie sweetener (LCS) consumption may affect this signaling in people with obesity. The aims will determine the independent and combined contributions of pharmacological inhibition (Aim 1) or extra stimulation (Aim 2) of sweet taste signaling in the gut, mouth, or both on hormonal responses to an oral glucose tolerance test (OGTT) in two groups of subjects with obesity: habitual and non-habitual LCS consumers. Validated sensory evaluation techniques will also ascertain subjects' taste perception (Aim 3) to test the hypotheses that habitual consumption of LCS blunts perception of sweetness and, in turn, affects postprandial glucose regulation.

ELIGIBILITY:
Inclusion Criteria:

* All races/ethnicities
* Habitual (> 5 diet sodas per week) and non-habitual (≤1 diet soda or 1 packet of LCS per week) LCS consumers
* 30 ≤ BMI <40 kg/m2
* Not severely insulin resistant (HOMA-IR2 < 2.6)

Exclusion Criteria:

* BMI < 30 and 40< BMI kg/m2
* HOMA-IR2>2.6
* Irregular LCS consumers (>1 diet sodas or packets of LCS per week but <5)
* Current smokers or quit smoking nicotine cigarettes for less than 6 months ago
* Pregnant, breastfeeding, menopausal
* Presence of anemia : <12g/dl for women and <13g/dl for men
* Blood donation in the past 8 weeks
* Presence of malabsorption syndrome
* History of bariatric surgery
* Presence of inflammatory intestinal disease, liver or kidney disease
* Have diabetes (fasting glucose level >126mg/dl or plasma glucose level 2h after glucose challenge >200 mg/dl)
* Taking any medication that might affect glucose metabolism or the results of our study

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma Glucose | Up to 5 hours after drinking a glucose load
  Blood samples will be collected before and for 5 hours after drinking a glucose load to determine plasma glucose concentration
Plasma Insulin | Up to 5 hours after drinking a glucose load
  Blood samples will be collected before and for 5 hours after drinking a glucose load to determine plasma insulin concentration
Plasma C-Peptide | Up to 5 hours after drinking a glucose load
  Blood samples will be collected before and for 5 hours after drinking a glucose load to determine plasma C-peptide concentration
Sensory Evaluation | Up to 2 hours
  Participants will be tasting solutions containing different concentrations of glucose, sucrose and sucralose (some of the solutions will also have lactisole) to assess their detection threshold, sweet taste intensity and preference. They will have to rate the intensity of the solution on a general Labeled Magnitude Scale (gLMS) ranging from "no sensation" (0) to "strongest imaginable sensation" (100) and choose the solutions they prefer.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana Champaign, Champaign, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the need to not compromise human subject protections, raw data that identifies participants will not be shared with anyone not included on our IRB approval. De-identified data, from participants who consented to share their de-identified data will be deposit in a data repository (e.g. Figshare).
Supporting Information: Study Protocol, ICF
Time Frame: We plan to share data no later than 6 months post-publication or 18 months from the award end date per ADA expectations.
Access Criteria: Data will be available to qualified individuals within the scientific community for research purposes contingent upon IRB approval for secondary data analysis.

REFERENCES:
- [Background] Adams TB, Cohen SM, Doull J, Feron VJ, Goodman JI, Marnett LJ, Munro IC, Portoghese PS, Smith RL, Waddell WJ, Wagner BM; Expert Panel of the Flavor and Extract Manufacturers Association. The FEMA GRAS assessment of phenethyl alcohol, aldehyde, acid, and related acetals and esters used as flavor ingredients. Food Chem Toxicol. 2005 Aug;43(8):1179-206. doi: 10.1016/j.fct.2004.11.013. Epub 2005 Jan 26. PMID 15950814
- [Background] Schiffman SS, Booth BJ, Sattely-Miller EA, Graham BG, Gibes KM. Selective inhibition of sweetness by the sodium salt of +/-2-(4-methoxyphenoxy)propanoic acid. Chem Senses. 1999 Aug;24(4):439-47. doi: 10.1093/chemse/24.4.439. PMID 10480680
- [Background] Jiang P, Cui M, Zhao B, Liu Z, Snyder LA, Benard LM, Osman R, Margolskee RF, Max M. Lactisole interacts with the transmembrane domains of human T1R3 to inhibit sweet taste. J Biol Chem. 2005 Apr 15;280(15):15238-46. doi: 10.1074/jbc.M414287200. Epub 2005 Jan 24. PMID 15668251
- [Background] Karimian Azari E, Smith KR, Yi F, Osborne TF, Bizzotto R, Mari A, Pratley RE, Kyriazis GA. Inhibition of sweet chemosensory receptors alters insulin responses during glucose ingestion in healthy adults: a randomized crossover interventional study. Am J Clin Nutr. 2017 Apr;105(4):1001-1009. doi: 10.3945/ajcn.116.146001. Epub 2017 Mar 1. PMID 28251932
- [Background] Pepino MY, Tiemann CD, Patterson BW, Wice BM, Klein S. Sucralose affects glycemic and hormonal responses to an oral glucose load. Diabetes Care. 2013 Sep;36(9):2530-5. doi: 10.2337/dc12-2221. Epub 2013 Apr 30. PMID 23633524
- [Background] Steinert RE, Gerspach AC, Gutmann H, Asarian L, Drewe J, Beglinger C. The functional involvement of gut-expressed sweet taste receptors in glucose-stimulated secretion of glucagon-like peptide-1 (GLP-1) and peptide YY (PYY). Clin Nutr. 2011 Aug;30(4):524-32. doi: 10.1016/j.clnu.2011.01.007. Epub 2011 Feb 15. PMID 21324568